CLINICAL TRIAL: NCT06890910
Title: Effect of Evidence Based Intervention on Sleep Quality Among Obese Pregnant Women:A Randomized Controlled Trial
Brief Title: Evidence Based Intervention for Improving Sleep Quality Among Obese Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Yehia Ali Mohamed, Lecturer of community health nursing at faculty of nursing/Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mohamed yehia Ali
Record Dates: First submitted 2025-03-15; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Sleep Disorders; Obese Pregnant Women
Keywords: sleep disorders, obesity, pregnant women, evidence based intervention
MeSH Terms: conditions — Sleep Wake Disorders; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: evidence based intervention
- control group (No Intervention)

INTERVENTIONS:
Other: evidence based intervention — sleep hygiene education. This education focused on four main aspects as follows:
  * Personal habits: Women were educated on establishing a regular bedtime routine, engaging in regular exercise, maintaining a healthy diet, avoiding caffeine and nicotine before bedtime, consuming adequate calcium and magnesium, drinking warm milk before sleep, and avoiding gas-producing foods or excessive fluid intake before bed.
  * Sleep environment: Women were advised to associate the bedroom only with sleep and intimacy, remove electronic devices, maintain a dark, quiet, and cool environment, ensure mattress and pillows were comfortable, and eliminate noise disturbances such as television.
  * Stimulus control: Participants were instructed to use the bed only for sleeping, avoid staying in bed if unable to sleep, and engage in minimally stimulating activities instead of worrying about insomnia.
  * Progressive muscle relaxation: Women in the study group received an educational session on the Jacobson's met
  Arms: study group

SUMMARY:
Sleep is essential for maternal and fetal health, with adequate sleep being crucial for energy, fetal development, and overall pregnancy well-being. However, sleep disturbances such as insomnia, sleep-disordered breathing (SDB), and restless legs syndrome (RLS) affect up to 83.5% of pregnant women, especially in the third trimester. These disturbances are linked to hormonal, anatomical, physiological, and psychological changes during pregnancy, as well as conditions like obesity, gestational hypertension, and gestational diabetes mellitus (GDM). Poor sleep quality can lead to cognitive impairment, fatigue, and increased risks for pregnancy complications, yet sleep disorders are often overlooked in prenatal care.

Obesity further exacerbates sleep disturbances, as excessive weight gain impacts endocrine pathways, increasing the risk of obstructive sleep apnea (OSA) and poor sleep quality. Research highlights the importance of good sleep hygiene, which includes a controlled sleep environment, dietary adjustments, and relaxation techniques such as progressive muscle relaxation (PMR). Behavioral therapies like relaxation exercises have shown promise in improving sleep, but there is limited high-quality research on their effectiveness during pregnancy.

Significance of the Study

Given the high prevalence of sleep disturbances in pregnancy and their potential negative effects on maternal and neonatal outcomes, this study aims to evaluate the impact of evidence-based interventions on sleep quality in obese pregnant women. Sleep disorders during pregnancy are associated with an increased risk of GDM, hypertension, cardiometabolic disorders, and postpartum depression. Effective interventions, such as sleep hygiene education and relaxation techniques, are cost-effective, feasible, and can be integrated into routine prenatal care. This study will contribute to evidence-based guidelines that could improve sleep health in pregnancy, benefiting both maternal and fetal well-being.

Aim & Hypothesis

The study aims to assess the effectiveness of evidence-based interventions in improving sleep quality among obese pregnant women through a randomized controlled trial (RCT). It hypothesizes that obese pregnant women receiving the intervention will demonstrate better sleep quality than those receiving routine antenatal care.

Methods

A parallel-group, open-label RCT was conducted in the antenatal clinic of Cairo University Hospitals. A total of 100 pregnant women meeting the eligibility criteria (BMI ≥30, gestational age 28-34 weeks, presence of sleep disturbance) were randomly assigned to either the intervention group (n=50) or control group (n=50). Exclusion criteria included high-risk pregnancies, known fetal abnormalities, preexisting psychiatric conditions, or prior treatment for sleep disorders.

Data Collection Tools:

Structured Interview Schedule - Collected demographic and obstetric history. Global Sleep Assessment Questionnaire (GSAQ) - Screened for sleep disturbances. Pittsburgh Sleep Quality Index (PSQI) - Assessed overall sleep quality. Sleep Hygiene Index (SHI) - Evaluated sleep habits. Intervention

Study Group: Received sleep hygiene education and relaxation training, including:

Personal habits (consistent sleep schedule, dietary adjustments, avoiding caffeine, using warm milk).

Sleep environment modifications (comfortable bed, removing electronic devices, noise control).

Stimulus control (associating the bed with sleep only, engaging in relaxation activities if unable to sleep).

Progressive Muscle Relaxation (PMR): Participants were trained in a structured relaxation technique, guided through video demonstrations, and given a handbook. They were instructed to practice PMR twice daily for four weeks.

Control Group: Received routine antenatal care, including general pregnancy monitoring without additional sleep-focused interventions.

Follow-up & Monitoring

Participants in the intervention group were followed up weekly via phone calls to ensure adherence to the interventions. Both groups underwent reassessments after four weeks using the same sleep evaluation tools.

Outcome Measures

Primary Outcome: Improved sleep quality (measured by PSQI) and Improved sleep hygiene (measured by SH .

Secondary Outcome:

ELIGIBILITY:
Inclusion Criteria:

* primigravida or multigravida women with any type of sleep disorder during pregnancy either insomnia, obstructive sleep apnea, restless leg syndrome, parasomnias; age 18-40 years old; obese women with body mass index (BMI) ≥ 30; being in the third trimester of pregnancy(28-34weeks of gestation)

Exclusion Criteria:

* having known risk of current pregnancy (preeclampsia, diabetes, heart disease, placenta previa, oligohydramnios, twin pregnancy, etc.); having known problem about fetus health (IUGR, anomaly, etc.); diagnosed with a sleep disorder for a different reasons and received treatment for it; history of psychiatric or somatic disorders; recent administration of psychoactive, sedative, or narcotic medications, and use of caffeine ( more than 8cups of coffee or 16 cups of tea/day).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
sleep quality | four weeks after intervention
  this outcome was assessed using Pittsburgh Sleep Quality Index (PSQI) . The PSQI is acommon method of examining the quality of sleep during pregnancy. The questionnaire includes seven components. These components include subjective sleep quality, sleep duration, sleep latency, sleep disturbances, the use of sleeping medication, daytime dysfunction habits and sleep efficiency.Each item is rated on a 0-3 scale, (zero) indicate very good, (1) indicate good,(2) indicate bad, and (3) indicate very bad.The sum of seven component scores gives the global PSQI score between 0 and 21. Ascore (0-4) indicated good sleep quality,score (5-10) indicated moderate sleep quality and score (11-21) indicated good sleep quality. The Cronbach's alpha of this questionnaire was calculated to be (0.83)
sleep hygiene | four weeks after intervention
  sleep hygiene was assessed using Sleep Hygiene Index (SHI). The tool was used as a self- report questionnaire, which can measure sleep hygiene. Sleep hygiene index has 13 items asking about sleeping habits as long naps , inconsistent bedtime ,inconsistent wake time ,late-night exercise , excessive time in bed ,substance use before bed ,stimulating activities before bed ,going to bed stressed ,using bed for non-sleep activities, uncomfortable bed, uncomfortable bedroom environment ,doing work before bed ,overthinking in bed. rating on a scale from 0 (never) to 4 (always). The global assessment score of SHI ranges from 0-52. Higher scores of SHI (score ≥ 16) indicate poor sleep hygiene and lower than 16 indicate good sleep hygiene. The reliability of the questionnaire was estimated to be(0.83)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of nursing at Cairo university, Cairo, Kase AlAini/El-Manial, Egypt